CLINICAL TRIAL: NCT06905301
Title: Implementation Study to Describe and Compare Retention Rate and Adherence to Adjuvant Therapy With Ribociclib With and Without Usage of Mobile Application in Patients With HR+ HER2-negative Stage II and III Breast Cancer in Real-world Practice
Acronym: IMPULSE
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLEE011O1RU01
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer
Keywords: Breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — ribociclib; Letrozole; Anastrozole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Using Application: HR + HER2- BC patients receiving adjuvant ribociclib + AI therapy in routine clinical practice that use the web application
  Interventions: Drug: Ribociclib; Drug: Letrozole; Drug: Anastrozole
- Non using Application: HR + HER2- BC patients receiving adjuvant ribociclib + AI therapy in routine clinical practice that do not use the web application
  Interventions: Drug: Ribociclib; Drug: Letrozole; Drug: Anastrozole

INTERVENTIONS:
Drug: Ribociclib — CDK4/6 inhibitor
Drug: Letrozole — Aromatase inhibitor
Drug: Anastrozole — Aromatase inhibitor

SUMMARY:
This study is designed to evaluate the effect of using the application on the adherence of patients with luminal HER2- breast cancer (BC) stage II-III to adjuvant therapy with ribociclib in combination with an aromatase inhibitor (AI). The purpose of the app is to increase adherence to treatment by informing patients about the risks of relapse and adverse event prevention and treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Female and male patients with histologically verified and radically treated stage II-III hormone receptor positive HER2-negative breast cancer;
2. Age ≥ 18 at the time of initiation of ribociclib therapy;
3. Patients who were prescribed ribociclib + AI (±GnRH agonist for premenopausal men and women) not earlier than 28 days before signing the informed consent;
4. It is allowed to start adjuvant hormone therapy with AI (±GnRH agonist) not earlier than 12 months before the start of ribociclib;
5. Provision of written informed consent.

Exclusion Criteria:

1. Patients participating in any interventional clinical study at the time of signing the informed consent;
2. Patients receiving active treatment for malignant neoplasms other than BC at the time of enrollment.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HR+ HER2- stage II-III breast cancer who have started treatment with ribociclib + AI (± GnRH agonist for premenopausal men and women) will be enrolled in the study
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2026-01-21 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Number (%) of patients who remain on treatment with ribociclib + AI over the 12 months period | 12 months
  The difference between the two groups (App and non-App) in number (%) of patients who remain on treatment with ribociclib + AI over the 12 months period (excluding patients who discontinued treatment due to AE, disease relapse, or death)

SECONDARY OUTCOMES:
Number of sessions using the web application per month | Month 1 - Month 36
  To describe the rate of the web application usage in the group of patients who use the web application.
Total duration of sessions (in minutes) per month | Month 1 - Month 36
  To describe the rate of the web application usage in the group of patients who use the web application.
Number of questions to the chatbot per month | Month 1 - Month 36
  To describe the rate of the web application usage in the group of patients who use the web application.
Evaluation of patient satisfaction with the application on a 0-10 visual analog scale (VAS) | Month 1, 3, 6, 12, 24, 36
  Evaluation of patient satisfaction with the application on a 0-10 VAS, where 0 is for completely dissatisfied, 10 is for completely satisfied in M1, M3, M6, M12, M24, M36
Evaluation of oncologist satisfaction with the application according to a 0-10 VAS | Month 1, 3, 6, 12, 24, 36
  Evaluation of oncologist satisfaction with the application according to a 0-10 VAS, where 0 is for completely dissatisfied, 10 is for completely satisfied in M1, M3, M6, M12, M24, M36
Number of patients in each response category according to the questionnaire on quality of life | Month 1, 3, 6, 12, 24, 36
  The number (%) of patients in each response category (no problems, mild problems, moderate problems, severe problems, and extremely severe problems) according to the questionnaire scale (mobility, self-care, normal activities, pain/discomfort, anxiety/depression) in M1, M3, M6, M12, M24, M36 in the groups using and not using the web application
VAS score according to the questionnaire on quality of life | Month 1, 3, 6, 12, 24, 36
  VAS score according to the questionnaire (VAS 0-100, where 0 is the worst health state and 100 is the best health state) at M1, M3, M6, M12, M24, and M36 in both app user and non-app user groups
Assessment of patient satisfaction with treatment | Month 3, 6, 12, 24, 36
  Assessment of patient satisfaction with treatment (VAS 0-10, where 0 is completely dissatisfied, and 10 is completely satisfied) at M3, M6, M12, M24, and M36 in both app user and non-app user groups
Dose intensity | Month 3, 6, 12, 24, 36
  Dose intensity (% of missed doses as assessed by the patient, except for therapy suspension due to AE) at M3, M6, M12, M24, and M36 in both app user and non-app user groups
Number of patients with adverse events (AE) | Month 3, 6, 12, 24, 36
  The percentage (%) of patients with AE (cumulative and depending on the severity) at M3, M6, M12, M24, and M36 in both app user and non-app user groups
Number of patients with dose reduction and/or discontinuation of ribociclib therapy due to progression, death for breast cancer, death from another cause, other AE | Month 3, 6, 12, 24, 36
  The percentage (%) of patients with dose reduction and/or discontinuation of ribociclib therapy due to progression, death for breast cancer, death from another cause, other AE at M3, M6, M12, M24, and M36 in both app user and non-app user groups
Number of patients by age, education, occupation, TNM (tumor, nodus, metastasis) stage, tumor grade (G), Ki67 level in both app user and non-app user groups | Baseline
  Proportion (%) of patients by age, education, occupation, TNM (tumor, nodus, metastasis) stage, tumor grade (G), Ki67 level in both app user and non-app user groups

CONTACTS AND LOCATIONS:
Locations (3):
- Russia (3):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Ufa